CLINICAL TRIAL: NCT05711615
Title: A Phase 1 Study of Peposertib (M3814) and Low-Dose Liposomal Doxorubicin in Patients With Metastatic Leiomyosarcoma and Other Soft Tissue Sarcomas
Brief Title: Testing Low-Dose Common Chemotherapy (Liposomal Doxorubicin) in Combination With an Anti-Cancer Drug, Peposertib, in Advanced Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-00574; NCI-2023-00574 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10563 (Other: Dana-Farber - Harvard Cancer Center LAO); 10563 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Dedifferentiated Liposarcoma; Metastatic Leiomyosarcoma; Metastatic Myxofibrosarcoma; Metastatic Sarcoma; Metastatic Synovial Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Unresectable Dedifferentiated Liposarcoma; Unresectable Leiomyosarcoma; Unresectable Myxofibrosarcoma; Unresectable Sarcoma; Unresectable Synovial Sarcoma; Unresectable Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Dermatofibrosarcoma; Sarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; liposomal doxorubicin; Doxorubicin; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (peposertib, liposomal doxorubicin) (Experimental): Patients receive peposertib PO BID on days 1-28 of each cycle and liposomal doxorubicin IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression, unacceptable toxicity or withdrawal of consent. Patients undergo blood sample collection and CT or MRI throughout the trial. Patients also undergo tissue biopsy and ECHO or MUGA during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Peposertib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Doxorubicin Liposomal; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of combination therapy with liposomal doxorubicin and peposertib in treating patients with sarcoma that has spread from where it first started, to other places in the body (metastatic), or cannot be removed by surgery (unresectable) and for which no known cure is available (advanced). Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's deoxyribonucleic acid (DNA) and may kill cancer cells. It also blocks a certain enzyme needed for cell division and DNA repair. Liposomal doxorubicin is a form of the anticancer drug doxorubicin that is contained inside very tiny, fat-like particles. Liposomal doxorubicin may have fewer side effects and work better than other forms of the drug. Peposertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also enhance the activity of chemo- and radiotherapy. There is some pre-clinical evidence in animal models that combining peposertib with liposomal doxorubicin can shrink or stabilize certain types of cancer for longer than either drug alone, but it is not known if this will happen in people. Combination therapy with liposomal doxorubicin and peposertib may be effective in treating patients with advanced sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of peposertib in combination with low-dose pegylated liposomal doxorubicin hydrochloride (liposomal doxorubicin) as evaluated by the dose-limiting toxicity (DLT) rate at each tested dose level. (Dose Escalation) II. To determine the recommended phase 2 dose (RP2D) of liposomal doxorubicin and peposertib combination and determine the maximal tolerated dose (MTD) if identified. (Dose Escalation) III. To obtain a more precise determination of adverse events (e.g. dose limiting toxicities estimate at the selected dose). (Dose Expansion)

SECONDARY OBJECTIVES:

I. To assess the pharmacokinetics of peposertib and liposomal doxorubicin used in combination with each other. (Dose Escalation) II. To estimate the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in patients with leiomyosarcoma treated with peposertib and low-dose liposomal doxorubicin. (Dose Expansion) III. To estimate the progression free survival (PFS) in patients with leiomyosarcoma treated with peposertib and low-dose liposomal doxorubicin. (Dose Expansion) IV. To assess the pharmacokinetics of peposertib and liposomal doxorubicin used in combination with each other. (Dose Expansion) V. To assess whether DNA damage is exaggerated by the low-dose liposomal doxorubicin in combination with peposertib in patients with homologous recombination (HR)-deficiency. (Dose Expansion)

CORRELATIVE OBJECTIVES:

I. To test the hypothesis that soft tissue sarcomas (STS) with homologous recombination deficiency (HRD) like leiomyosarcomas (LMS) will be more susceptible to DNA-protein kinase inhibitor (PKi) in combination with low-dose liposomal doxorubicin.

II. To test the hypothesis that gammaH2AX and pNBS1 can be used as pharmacodynamic biomarkers of response to DNA-PKi in combination with low-dose liposomal doxorubicin.

III. To test the hypothesis that disease activity correlates with circulating tumor DNA levels in the plasma.

OUTLINE: This is a dose-escalation study of peposertib and liposomal doxorubicin followed by a dose-expansion study.

Patients receive peposertib orally (PO) twice daily (BID) on days 1-28 of each cycle and liposomal doxorubicin intravenously (IV) on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression, unacceptable toxicity or withdrawal of consent. Patients undergo blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients also undergo tissue biopsy and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and on the trial.

Patients are followed for 30 days after removal from study or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed sarcoma that is metastatic or unresectable and for which there is no known curative treatment
* Dose escalation cohort: Patients must have histologic diagnosis of leiomyosarcoma (LMS) or selected soft tissue sarcomas (myxofibrosarcoma [MFS], undifferentiated pleomorphic sarcoma [UPS], synovial sarcoma, or dedifferentiated liposarcoma [DDLPS]). Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study
* Dose expansion cohort: Patients must have histology diagnosis of LMS. Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study
* Dose escalation cohort: Patients must have evaluable disease that is amenable to biopsy
* Dose expansion cohort: Patients must have disease which is measurable at study entry according to RECIST 1.1 criteria and amenable to biopsy
* Patients must have been treated with at least 1 prior line of therapy. Prior anthracycline use is permitted as long as the cumulative dose prior to enrollment does not exceed 360 mg/m^2
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of peposertib (M3814) in combination with liposomal doxorubicin in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%) for both dose escalation and dose expansion
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Hemoglobin >= 8 g/dL
* Glomerular filtration rate (GFR) >= 51 mL/min/1.73 m^2 (per institutional estimate based on creatinine level)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and clinical symptoms are stable while off steroid support
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history of clinically significant cardiac disease, or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 3 months after the last dose of peposertib (M3814) and 6 months after the last dose of liposomal doxorubicin
* Male patients of reproductive potential must agree to avoid impregnating a partner while receiving study drug and for 3 months after the last dose of peposertib (M3814) and 6 months after the last dose of liposomal doxorubicin by complying with adequate methods of contraception

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Prior palliative radiotherapy within 14 days of cycle 1 day 1 and prior definitive radiotherapy within 42 days of cycle 1 day 1. Adverse effects of radiation therapy must resolve to baseline prior to cycle 1 day 1
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to peposertib (M3814) or other agents used in study
* Patients who cannot discontinue concomitant medications or herbal supplements that are strong inhibitors or strong inducers of cytochrome P450 (CYP) isoenzymes CYP3A4/5, CYP2C9, and CYP2C19. Participants who cannot discontinue substrates with a narrow therapeutic index that are metabolized by CYP1A2, CYP2B6, CYP2C8, and CYP3A4/5 are ineligible. Patients may confer with the study doctor to determine if alternative medications can be used. The following categories of medications and herbal supplements must be discontinued for at least the specified period of time before the patient can be treated:

  * Strong inducers of CYP3A4/5 and CYP2C19: >= 3 weeks prior to study treatment
  * Strong inhibitors of CYP3A4/5 and CYP2C19: >= 1 week prior to study treatment
  * Substrates of CYP3A4/5 with a narrow therapeutic index: >= 1 day prior to study treatment
  * Strong inhibitors of CYP2C9: >= 1 week prior to study treatment
* Patients who cannot discontinue concomitant proton-pump inhibitors (PPIs). Patients may confer with the study doctor to determine if such medications can be discontinued. These must be discontinued >= 5 days prior to study treatment. Patients do not need to discontinue calcium carbonate
* Patients with left ventricular ejection fraction (LVEF) measurement below the institutional lower limit of normal (LLN) are excluded
* Patients with uncontrolled intercurrent illness
* Patients who cannot swallow tablets whole
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are not eligible
* Pregnant women are excluded from this study because peposertib (M3814) is an adenosine triphosphate (ATP)-competitive inhibitor of DNA-protein kinase catalytic subunit (PKcs) with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with peposertib (M3814), breastfeeding should be discontinued if the mother is treated with peposertib (M3814). These potential risks may also apply to other agents used in this study
* Patients may not have received prior treatment with a DNA-protein kinase (PK) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | Up to 28 days
  The number and type of DLT seen at each dose level will be provided. The adverse events (AEs) will also be summarized by AE type and the maximum grade of the AE experienced by the patient for each dose level. DLT will be used to determine the recommended phase 2 dose of study drugs.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the end of study treatment
  AEs will be assessed using Common Terminology Criteria for Adverse Events version 5.
Objective response rate | Up to 28 days
  Assessed with Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.
Progression free survival | From study enrollment until disease progression (determined by RECIST v1.1) or death due to any cause, whichever occurs first
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. Patients who are alive at the time of analysis without a documented disease progression will be censored at the time of their last tumor evaluation.
Homologous recombination deficiency (HRD) status | Up to 1 year
  Will be defined by HRD score and mutational signature analysis.
Deoxyribonucleic acid damage repair activity | Up to 1 year
  Will be defined by gammaH2AX and NBS1 S343 phosphorylation based on the National Clinical Laboratory Network DDR3 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Candace L Haddox, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (16):
- United States (16):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm